CLINICAL TRIAL: NCT06427538
Title: Chest Drain Regular Flushing in Complicated Parapneumonic Effusions and Empyemas
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Samira Shojaee, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 231367
Record Dates: First submitted 2024-05-10; First posted 2024-05-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Empyema, Pleural; Pleural Infection
Keywords: empyema; pleural infection; chest tube; saline flush
MeSH Terms: conditions — Empyema, Pleural; Empyema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline Intervention Arm (Experimental): Patient will receive 20 mL sterile saline flushes into their catheter by study team members every 6 ± 2 hours. If patients are receiving intrapleural tissue plasminogen activator and deoxyribonuclease therapy, each treatment will be considered one flush.
  Interventions: Other: Saline Flush
- No Intervention Arm (No Intervention): Patient will receive a saline flush as needed, to restore patency of a chest tube considered blocked. No routine flushes will be administered.

INTERVENTIONS:
Other: Saline Flush — sterile saline 20 mL flushed into their catheter by trained nurses or study team members every 6 ± 2 hours
  Arms: Saline Intervention Arm

SUMMARY:
Infections of the pleural space are common, and patients require antibiotics and chest drain placement to evacuate the chest from the infected fluid. Chest drains can get blocked by the drainage fluid and material. For this reason, it is thought that flushing the chest drain with saline solution, can help maintain the patency of the tube. This proposed study will evaluate the impact of regular chest drain flushing on the length of time to chest tube removal and total hospitalization as well as improvement in chest imaging and the need for additional interventions on the infected space.

DETAILED DESCRIPTION:
There are no randomized controlled trials (RCTs) evaluating the role of regular chest tube flushing in the setting of pleural space infection for optimal drainage and treatment outcomes. Most studies of <16 Fr catheters have used both flushing and suction to decrease the likelihood of catheter blockage and improve drainage efficiency, however, this practice has never been studied prospectively or in RCTs. Regular flushing (e.g., 20-30 ml saline every 6 h via a three-way tap) is recommended for small chest drains by the British Thoracic Society (BTS) 2010 Guidelines. This practice is followed variably by some and not used by others. Importantly, the role of this practice in successful drainage of infected fluid, and patient-centric outcomes has not been investigated. Inconsistent flushing practices confound the interpretation of therapeutic modalities (such as intrapleural tissue plasminogen activator and deoxyribonuclease therapy) success or lack thereof and limit the execution of RCTs and prospective studies of the pleural space in the setting of infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complicated parapneumonic pleural effusion and empyema requiring chest tube placement as standard of care for inpatient management of their pleural space infection with or without intrapleural tissue plasminogen activator and deoxyribonuclease therapy
* Age > 18 years old.

Exclusion Criteria:

* Patients who have surgical tubes that can't accommodate a three-way stopcock.
* Study subject has any disease or condition that interferes with the safe completion of the study.
* Inability to provide informed consent.
* Inability to undergo a chest X-ray.
* If the managing clinician believes the chest tube will be placed for less than 24 hours.
* Patients with an indwelling pleural catheter (IPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Time to chest tube removal | up to 3 months
  The investigators will assess the time from randomization (within 24 hours of chest tube placement) until time to chest tube removal

SECONDARY OUTCOMES:
Length of hospitalization | up to 365 days
Radiographic improvement as evidenced by chest x-ray at the time of chest tube placement compared to the time of removal | through study completion, an average of 3 months
Additional surgical procedures for the management of pleural space infection | an average of 3 months
  number of additional procedures through study completion
Complications | through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Duke, MD, Study Director — Vanderbilt University
Locations (5):
- United States (5):
  - Henry Ford, Sterling Heights, Michigan
  - Creighton University, Omaha, Nebraska
  - Mount Sinai, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared with other researchers